CLINICAL TRIAL: NCT04288115
Title: Discontinuation of Levothyroxine Therapy for Patients With Subclinical Hypothyroidism: a Pilot Randomized, Double-blinded, Placebo-controlled Study
Brief Title: Discontinuation of Levothyroxine Therapy for Patients With Subclinical Hypothyroidism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Central Arkansas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PPO 20-056; 1521422 (Other Grant/Funding Number: Central Arkansas Veterans Healthcare System)
Record Dates: First submitted 2020-02-14; First posted 2020-02-28 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Subclinical Hypothyroidism
MeSH Terms: interventions — Thyroxine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Levothyroxine group ("sham discontinuation") (Active Comparator): Continue the current dose of levothyroxine. The brand of levothyroxine to be used in this study will be Synthroid tablets of 25 mcg, 50 mcg, and 75 mcg (AbbVie Inc).
  Interventions: Drug: Levothyroxine
- Placebo group ("real discontinuation") (Placebo Comparator): Stop the current dose of levothyroxine and take study placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Levothyroxine — Participants will be instructed to start the study medication the day after randomization. The study medication will be taken orally once a day.
  Other Names: Synthroid
  Arms: Levothyroxine group ("sham discontinuation")
Other: Placebo — Participants will be instructed to start the study medication the day after randomization. The study medication will be taken orally once a day.
  Arms: Placebo group ("real discontinuation")

SUMMARY:
The investigators propose the following hypothesis: discontinuation of levothyroxine (LT4) for veterans with subclinical hypothyroidism (SCH) will be feasible, acceptable, and safe and will not negatively affect their Quality of Life (QoL). The investigators aim to evaluate the feasibility of LT4 discontinuation among veterans with SCH and determine the changes in QoL measures, lipids, and adverse events.

DETAILED DESCRIPTION:
This is a pilot, randomized, double-blind, placebo-controlled trial.

Methodology:

The investigators will conduct a double-blind, placebo-controlled clinical trial where eligible veterans diagnosed with SCH and on LT4 will be 1:1 randomized to either continue LT4 or change to placebo. The primary outcome is intervention feasibility (willingness to enter the trial, recruitment rate, and completion rate). Secondary outcomes are: 1) changes in QoL measures (Hypothyroid Symptom [HSS] and Tiredness scale scores of the Thyroid-Specific Patient-Related Outcome Measure [ThyPRO], EuroQoL 5-Dimension Self-Report Questionnaire) measured at baseline, 6-8 weeks and 6 months and 2) changes in lipids assessed at baseline and 6 months, and 3) incidence of adverse events (overt hypothyroidism, hyperthyroidism, atrial fibrillation, fractures, acute myocardial infarction, stroke, acute coronary syndrome, heart failure, mortality).

ELIGIBILITY:
Inclusion Criteria:

* Veterans
* diagnosis of SCH

Exclusion Criteria:

* thyroid-stimulating hormone (TSH) > 10 milli-international units per liter (mlU/L) (at any point)
* Levothyroxine (LT4) dose more than 75 mcg daily
* use of antithyroid medications, amiodarone, tyrosine kinase inhibitors or lithium
* history of thyroidectomy or radioactive iodine therapy
* LT4 suppressive therapy for thyroid cancer, goiter, or inflammation
* pregnancy or plans for pregnancy in the next 6 months
* an unstable medical condition that would jeopardize safety or interfere with study participation
* severe hypothyroidism-related symptoms
* strong family history of hypothyroidism
* severe dyslipidemia
* hospitalization for major illness within the previous 4 weeks
* acute coronary artery syndrome, acute myocarditis, or pancarditis with the previous 12 months
* grade IV New York Heart Association heart failure
* receiving services from hospice
* lack of decision-making capacity
* terminal medical condition for which life expectancy would be less than 6 months
* not willing to stop LT4
* self-reported non-adherence to LT4 therapy
* abnormal TSH at time of screening for participation (assessed during Baseline Visit)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Spyridoula Maraka, MD MS, Principal Investigator — Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR
Locations (1):
- Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR, North Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brito JP, Ross JS, El Kawkgi OM, Maraka S, Deng Y, Shah ND, Lipska KJ. Levothyroxine Use in the United States, 2008-2018. JAMA Intern Med. 2021 Oct 1;181(10):1402-1405. doi: 10.1001/jamainternmed.2021.2686. PMID 34152370
- [Background] Feller M, Snel M, Moutzouri E, Bauer DC, de Montmollin M, Aujesky D, Ford I, Gussekloo J, Kearney PM, Mooijaart S, Quinn T, Stott D, Westendorp R, Rodondi N, Dekkers OM. Association of Thyroid Hormone Therapy With Quality of Life and Thyroid-Related Symptoms in Patients With Subclinical Hypothyroidism: A Systematic Review and Meta-analysis. JAMA. 2018 Oct 2;320(13):1349-1359. doi: 10.1001/jama.2018.13770. PMID 30285179
- [Background] Stott DJ, Rodondi N, Kearney PM, Ford I, Westendorp RGJ, Mooijaart SP, Sattar N, Aubert CE, Aujesky D, Bauer DC, Baumgartner C, Blum MR, Browne JP, Byrne S, Collet TH, Dekkers OM, den Elzen WPJ, Du Puy RS, Ellis G, Feller M, Floriani C, Hendry K, Hurley C, Jukema JW, Kean S, Kelly M, Krebs D, Langhorne P, McCarthy G, McCarthy V, McConnachie A, McDade M, Messow M, O'Flynn A, O'Riordan D, Poortvliet RKE, Quinn TJ, Russell A, Sinnott C, Smit JWA, Van Dorland HA, Walsh KA, Walsh EK, Watt T, Wilson R, Gussekloo J; TRUST Study Group. Thyroid Hormone Therapy for Older Adults with Subclinical Hypothyroidism. N Engl J Med. 2017 Jun 29;376(26):2534-2544. doi: 10.1056/NEJMoa1603825. Epub 2017 Apr 3. PMID 28402245
- [Background] Bekkering GE, Agoritsas T, Lytvyn L, Heen AF, Feller M, Moutzouri E, Abdulazeem H, Aertgeerts B, Beecher D, Brito JP, Farhoumand PD, Singh Ospina N, Rodondi N, van Driel M, Wallace E, Snel M, Okwen PM, Siemieniuk R, Vandvik PO, Kuijpers T, Vermandere M. Thyroid hormones treatment for subclinical hypothyroidism: a clinical practice guideline. BMJ. 2019 May 14;365:l2006. doi: 10.1136/bmj.l2006. PMID 31088853
- [Background] Ayala IN, Soto Jacome C, Toro-Tobon D, Golembiewski E, Garcia-Bautista A, Hidalgo J, Cordova-Madera S, Al Anbari R, Sohn R J, Singh Ospina N, Maraka S, Joseph M, Brito JP. Appropriateness of Levothyroxine Prescription: A Multicenter Retrospective Study. J Clin Endocrinol Metab. 2024 Jan 18;109(2):e765-e772. doi: 10.1210/clinem/dgad517. PMID 37656124
- [Background] Toloza FJK, El Kawkgi OM, Spencer HJ, Mathews SE, Garcia A, Gamboa A, Mirza N, Mohan S, Vallejo S, Bogojevic M, Rodriguez-Gutierrez R, Singh Ospina NM, Brito JP, Maraka S. Determinants for Thyroid Hormone Replacement Therapy in Subclinical Hypothyroidism: A Multicenter Electronic Health Records-Based Study. Thyroid. 2023 Sep;33(9):1045-1054. doi: 10.1089/thy.2023.0062. Epub 2023 Jun 26. PMID 37279296
- [Background] Ospina NS, Salloum RG, Maraka S, Brito JP. De-implementing low-value care in endocrinology. Endocrine. 2021 Aug;73(2):292-300. doi: 10.1007/s12020-021-02732-y. Epub 2021 May 11. PMID 33977312
- [Background] Burgos N, Toloza FJK, Singh Ospina NM, Brito JP, Salloum RG, Hassett LC, Maraka S. Clinical Outcomes After Discontinuation of Thyroid Hormone Replacement: A Systematic Review and Meta-Analysis. Thyroid. 2021 May;31(5):740-751. doi: 10.1089/thy.2020.0679. Epub 2020 Dec 29. PMID 33161885
- [Derived] Maraka S, Owen RR, Singh Ospina NM, Knox M, Dodds T, Thostenson JD, Dishongh K, Raciborski RA, Albashaireh A, Shah A, Syed S, Naqvi S, Motahari H, Thumma S, Toloza F, Ambrogini E, Brito JP. Discontinuation of levothyroxine therapy in patients with subclinical hypothyroidism: a pilot randomized clinical trial. Endocrine. 2025 Nov;90(2):781-792. doi: 10.1007/s12020-025-04371-z. Epub 2025 Jul 30. PMID 40736623

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on opt-in/opt-out letter at 1 VA medical center between March 2021 and April 2022. The first participant was enrolled on March 24, 2021 and the last participant was enrolled in April 2022.
Pre-assignment Details: Of 52 enrolled participants, 50 were randomized to treatment.
Period: Overall Study
Arm/Group | Levothyroxine Group ("Sham Discontinuation") | Placebo Group ("Real Discontinuation")
Started | 24 | 26
Completed | 21 | 23
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Pre-study SCH diagnosis could not be confirmed per study entry criteria | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levothyroxine Group ("Sham Discontinuation") | Placebo Group ("Real Discontinuation") | Total
Number analyzed (Participants) | 21 | 24 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.0 (7.9) | 65.7 (10.6) | 68.2 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 18 | 18 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 21 | 23 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 18 | 21 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 24 | 45
Weight [Mean (Standard Deviation); unit: pounds] | 220.4 (58.4) | 201.0 (61.5) | 210.1 (60.2)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 32.5 (7.7) | 29.7 (7.8) | 31.0 (7.8)
Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: mm Hg] | 141.1 (19.7) | 137.5 (16.8) | 139.2 (18.1)
Diastolic Blood Pressure (DBP) [Mean (Standard Deviation); unit: mm Hg] | 80.1 (8.7) | 80.2 (11.7) | 80.1 (10.3)
Pulse [Mean (Standard Deviation); unit: beats/min] | 68.3 (15.7) | 66.8 (9.4) | 67.5 (12.6)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 148.1 (41.9) | 179.8 (31.3) | 165.0 (39.6)
LDL [Mean (Standard Deviation); unit: mg/dL] | 77.5 (34.5) | 104.2 (28.4) | 91.7 (33.9)
HDL [Mean (Standard Deviation); unit: mg/dL] | 42.4 (11.5) | 53.3 (19.8) | 48.2 (17.2)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] | 141.5 (68.0) | 111.4 (48.0) | 125.4 (59.5)
Levothyroxine (LT4) dose prior to enrollment, 25mcg [Count of Participants; unit: Participants] | 7 | 7 | 14
LT4 dose prior to enrollment, 50mcg [Count of Participants; unit: Participants] | 10 | 13 | 23
LT4 dose prior to enrollment, 75mcg [Count of Participants; unit: Participants] | 4 | 4 | 8
LT4 duration, < 2 yrs [Count of Participants; unit: Participants] | 6 | 6 | 12
LT4 duration, 2 to 7 yrs [Count of Participants; unit: Participants] | 10 | 12 | 22
LT4 duration, > 7 yrs [Count of Participants; unit: Participants] | 5 | 6 | 11
thyroid-stimulating hormone (TSH) [Mean (Standard Deviation); unit: mIU/L] | 3.19 (1.42) | 3.08 (0.99) | 3.1 (1.2)
free thyroxine (FT4) [Mean (Standard Deviation); unit: ng/dL] | 0.9 (0.1) | 0.9 (0.1) | 0.9 (0.1)
thyroid peroxidase (TPO) positivity [Count of Participants; unit: Participants] | 4 | 4 | 8
Hypothyroid Symptoms score [Mean (Standard Deviation); unit: scores on scale] — The Hypothyroid Symptoms score from the Thyroid-Related Quality of Life Patient-Reported Outcome (ThyPRO) questionnaire is assessed on a scale from 0 to 100, with higher scores indicating more symptoms. The minimum clinically important difference has been estimated as 9 points.
  scores on scale | 21.1 (18.4) | 27.1 (20.4) | 24.3 (19.5)
Tiredness score [Mean (Standard Deviation); unit: scores on scale] — The Tiredness score from the Thyroid-Related Quality of Life Patient-Reported Outcome (ThyPRO) questionnaire is assessed on a scale from 0 to 100, with higher scores indicating more tiredness. The minimum clinically important difference has been estimated as 9 points.
  scores on scale | 31.1 (23.9) | 33.2 (23.7) | 32.2 (23.5)
ThyPRO-39 score [Mean (Standard Deviation); unit: scores on scale] — ThyPRO-39 scales range 0-100, with higher levels corresponding to more symptoms or more quality of life impairment.
  scores on scale | 20.5 (14.8) | 18.4 (11.2) | 19.4 (12.9)
EQ-5D Descriptive score [Mean (Standard Deviation); unit: scores on scale] — The EuroQoL [EQ] Group 5-Dimension Self-Report Questionnaire (EQ-5D) scores include the EQ-5D descriptive index, on a scale from -0.59 to 1.00. Higher scores indicate better quality of life.
  scores on scale | 0.758 (0.193) | 0.746 (0.229) | 0.752 (0.210)
EQ-5D VAS score [Mean (Standard Deviation); unit: scores on scale] — The EuroQoL [EQ] Group 5-Dimension Self-Report Questionnaire (EQ-5D) scores include the score on the EQ visual-analogue scale (EQ-5D VAS), on a scale from 0 to 100. Higher scores indicate better quality of life.
  scores on scale | 72.0 (15.0) | 77.3 (14.4) | 74.8 (14.7)

OUTCOME MEASURES:

1. Primary Outcome: Participants' Willingness to Enter the Trial
Description: Percent of eligible participants approached who consented to participate during the recruitment phase.
Time Frame: The time from first consent signed to last consent signed. March 2021 to April 2022.
Population: The number of patients consented divided by the total number of eligible patients contacted.
Measure: Count of Participants; unit: Participants
Groups:
- Percentage of Eligible Patients Willing to Participate.: The percentage of eligible patients that were willing to participate and were enrolled (signed consent) from the total number of patients contacted.
Arm/Group | Percentage of Eligible Patients Willing to Participate.
Number analyzed (Participants) | 162
Participants | 52

2. Primary Outcome: Recruitment Rate
Description: The number of enrolled (consented) participants divided by the length of the recruitment period.
Time Frame: The time from first consent signed to last consent signed. March 2021 to April 2022. 13 months.
Population: The number of participants enrolled divided by the length of recruitment period (13 months).
Measure: Number; unit: participants per month
Groups:
- Recruitment Rate: A calculation of the recruitment rate of participant enrollment per month.
Arm/Group | Recruitment Rate
Number analyzed (Participants) | 52
participants per month | 4

3. Primary Outcome: Completion Rate
Description: Percentage of randomized participants who completed the trial.
Time Frame: 6 months
Population: Number of randomized participants that completed the trial divided by the total number of randomized participants.
Measure: Count of Participants; unit: Participants
Groups:
- Randomized Participants: Percentage of randomized participants who completed the trial.
Arm/Group | Randomized Participants
Number analyzed (Participants) | 45
Participants | 44

4. Secondary Outcome: Thyroid-specific Quality of Life Patient-Reported Outcome (ThyPRO) - Hypothyroid Symptoms Score
Description: The Hypothyroid Symptoms score from the Thyroid-Related Quality of Life Patient-Reported Outcome (ThyPRO) questionnaire is assessed on a scale from 0 to 100, with higher scores indicating more symptoms.
Time Frame: Baseline, 6 weeks and 6 months
Population: All randomized participants who completed 6 months follow-up visit. An intent-to-treat strategy was employed where participants were analyzed in the group to which they were randomized, regardless of protocol deviations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Levothyroxine Group ("Sham Discontinuation") | Placebo Group ("Real Discontinuation")
Number analyzed (Participants) | 21 | 23
score on a scale
  Baseline | 21.1 (18.4) | 27.1 (20.4)
  6 weeks | 22.0 (17.7) | 25.3 (21.9)
  6 months | 22.9 (19.5) | 28.3 (22.8)
Statistical Analysis 1: Comparison: Levothyroxine Group ("Sham Discontinuation") vs Placebo Group ("Real Discontinuation"); A one-sided t-test will be used to determine whether the mean Hypothyroid Symptoms score for the real discontinuation group is no more than 14 points worse than the score of the sham discontinuation group at 6 months; Test type: Non-Inferiority — An one-sided α-level of 0.05 will be used to determine the statistical significance of the non-inferiority test; p = 0.0913, Welch's two-sample t-test — Group differences; A one-sided p-value < 0.05 indicates the discontinuation mean falls within the non-inferiority limit; Difference in Group Means = -5.3, 90% CI 2-sided [-16.1 to 5.4] — Differences reported as the sham discontinuation mean minus the real discontinuation mean
Statistical Analysis 2: Comparison: Levothyroxine Group ("Sham Discontinuation") vs Placebo Group ("Real Discontinuation"); Analysis of 6-week outcome; Test type: Other — A two-sided α-level of 0.05 will be used to determine the statistical difference; p = 0.8793, ANCOVA — Testing whether group means are different; A p-value < 0.05 indicates the real discontinuation mean and the sham discontinuation mean are different. Adjusted for gender and baseline HSSs; Difference in Group Means = 0.8, 95% CI 2-sided [-9.4 to 10.9] — Differences reported as the sham discontinuation mean minus the real discontinuation mean. These differences have been adjusted for gender and baseline hypothyroid symptom scores
Statistical Analysis 3: Comparison: Levothyroxine Group ("Sham Discontinuation") vs Placebo Group ("Real Discontinuation"); Analysis of 6-month outcome; Test type: Other — A two-sided α-level of 0.05 will be used to determine the statistical significance; p = 0.6860, ANCOVA — Group differences; A p-value < 0.05 indicates real discontinuation mean and sham discontinuation mean are different. Analyses adjusted for gender and baseline HSS; Difference in Group Means = -2.3, 95% CI 2-sided [-14.0 to 9.3] — Differences are reported as sham discontinuation mean minus real discontinuation mean. These differences have been adjusted for gender and baseline hypothyroid symptom scores

5. Secondary Outcome: Thyroid-specific Quality of Life Patient-Reported Outcome (ThyPRO) - Tiredness Score
Description: The Tiredness score from the Thyroid-Related Quality of Life Patient-Reported Outcome (ThyPRO) questionnaire is assessed on a scale from 0 to 100, with higher scores indicating more tiredness.
Time Frame: Baseline, 6 weeks and 6 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Levothyroxine Group ("Sham Discontinuation") | Placebo Group ("Real Discontinuation")
Number analyzed (Participants) | 21 | 23
score on a scale
  Baseline | 31.1 (23.9) | 33.2 (23.7)
  6 weeks | 33.0 (23.6) | 31.1 (24.3)
  6 months | 32.8 (22.1) | 27.6 (22.8)
Statistical Analysis 1: Comparison: Levothyroxine Group ("Sham Discontinuation") vs Placebo Group ("Real Discontinuation"); A one-sided t-test will be used to determine whether the mean Tiredness score for the real discontinuation group is no more than 14 points worse than the score of the sham discontinuation group at 6 months; Test type: Non-Inferiority — A one-sided α-level of 0.05 will be used to determine the statistical significance of the non-inferiority test; p = 0.0036, Welch's two-sample t-test — Group differences; A one-sided p-value < 0.05 indicates the discontinuation mean falls within the non-inferiority limit; Difference in Group Means = 5.2, 90% CI 2-sided [-6.2 to 16.6] — Differences reported as the sham discontinuation mean minus the real discontinuation mean
Statistical Analysis 2: Comparison: Levothyroxine Group ("Sham Discontinuation") vs Placebo Group ("Real Discontinuation"); Analysis of 6-week outcome; Test type: Other — A two-sided α-level of 0.05 will be used to determine the statistical significance; p = 0.7104, ANCOVA — Testing whether group means are different; A p-value < 0.05 indicates real discontinuation mean and sham discontinuation mean are different. Analyses adjusted for gender and baseline score; Difference in Group Means = 2.3, 95% CI 2-sided [-10.1 to 14.7] — Differences reported as the sham discontinuation mean minus the real discontinuation mean. These mean differences have been adjusted for gender and baseline tiredness score
Statistical Analysis 3: Comparison: Levothyroxine Group ("Sham Discontinuation") vs Placebo Group ("Real Discontinuation"); Analysis of 6-month outcome; Test type: Other — A two-sided α-level of 0.05 will be used to determine statistical significance; p = 0.3381, ANCOVA — Group differences; [statistical method as in outcome 5, analysis 2]; Difference in Group Means = 5.4, 95% CI 2-sided [-5.9 to 16.7] — Differences reported as sham discontinuation mean minus real discontinuation mean. These differences have been adjusted for gender and baseline tiredness scores

6. Secondary Outcome: Euro Quality of Life 5-Dimension Self-Report Questionnaire (EQ-5D) Score at Week 6 and Month 6
Description: The EuroQoL [EQ] Group 5-Dimension Self-Report Questionnaire (EQ-5D) scores include the EQ-5D descriptive index, on a scale from -0.59 to 1.00. Higher scores indicate better quality of life. The EQ-5D scores include the score on the EQ visual-analogue scale (EQ-5D VAS), on a scale from 0 to 100. Higher scores indicate better quality of life.
Time Frame: 6 weeks and 6 months
Population: All randomized participants who completed 6 months follow-up visit. An intent-to-treat strategy was employed where participants were analyzed into the group they were randomized, regardless of protocol deviations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Levothyroxine Group ("Sham Discontinuation") | Placebo Group ("Real Discontinuation")
Number analyzed (Participants) | 21 | 23
score on a scale
  EQ-5D Descriptive Score 6 weeks | 0.759 (0.190) | 0.786 (0.214)
  EQ-5D Descriptive Score 6 months | 0.742 (0.180) | 0.750 (0.232)
  EQ-5D VAS 6 weeks | 78.0 (13.8) | 77.2 (19.6)
  EQ-5D VAS 6 months | 68.4 (21.2) | 79.9 (12.9)
Statistical Analysis 1: Comparison: Levothyroxine Group ("Sham Discontinuation") vs Placebo Group ("Real Discontinuation"); Analysis of 6-week EQ-5D Descriptive score outcome; Test type: Other — A two-sided α-level of 0.05 will be used to determine the statistical significance; p = 0.4684, ANCOVA — Testing whether group means are different; [statistical method as in outcome 5, analysis 2]; Difference in Group Means = -0.020, 95% CI 2-sided [-0.076 to 0.036] — Differences reported as the sham discontinuation mean minus the real discontinuation mean. These differences have been adjusted for gender and baseline EQ-5D Descriptive scores
Statistical Analysis 2: Comparison: Levothyroxine Group ("Sham Discontinuation") vs Placebo Group ("Real Discontinuation"); Analysis of 6-month EQ-5D Descriptive score outcome; Test type: Other — A two-sided α-level of 0.05 will be used to determine the statistical significance; p = 0.9585, ANCOVA — Testing whether group means are different; [statistical method as in outcome 5, analysis 2]; Difference in Group Means = 0.003, 95% CI 2-sided [-0.102 to 0.107] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Levothyroxine Group ("Sham Discontinuation") vs Placebo Group ("Real Discontinuation"); Analysis of 6-week EQ-5D VAS score outcome; Test type: Other — A two-sided α-level of 0.05 will be used to determine the statistical significance; p = 0.0643, ANCOVA — Testing whether group means are different; [statistical method as in outcome 5, analysis 2]; Difference in Group Means = 7.0, 95% CI 2-sided [-0.4 to 14.4] — Differences reported as the sham discontinuation mean minus the real discontinuation mean. These differences have been adjusted for gender and baseline EQ-5D VAS scores
Statistical Analysis 4: Comparison: Levothyroxine Group ("Sham Discontinuation") vs Placebo Group ("Real Discontinuation"); Analysis of 6-month EQ-5D VAS score outcome; Test type: Other — A two-sided α-level of 0.05 will be used to determine the statistical significance; p = 0.1742, ANCOVA — Testing whether group means are different; A p-value < 0.05 indicates real discontinuation mean and sham discontinuation mean are different. Analyses adjusted for gender and baseline scores; Difference in Group Means = -6.2, 95% CI 2-sided [-15.3 to 2.9] — [estimate comment as in outcome 6, analysis 3]

7. Secondary Outcome: Lipid Levels
Description: Differences in mean 6-month lipid levels after adjusting for gender and baseline lipid level.
Time Frame: 6 months
Population: All participants who completed 6-8 weeks and 6 months follow-up visit.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Levothyroxine Group ("Sham Discontinuation") | Placebo Group ("Real Discontinuation")
Number analyzed (Participants) | 21 | 23
mg/dL
  Total cholesterol 6 months | 145.3 (32.6) | 177.4 (39.6)
  LDL 6 months | 76.5 (28.6) | 100.2 (32.3)
  HDL 6 months | 42.7 (16.5) | 51.5 (16.2)
  Triglycerides 6 months | 137.5 (66.8) | 139.7 (68.4)
Statistical Analysis 1: Comparison: Levothyroxine Group ("Sham Discontinuation") vs Placebo Group ("Real Discontinuation"); Analysis of 6-month total cholesterol outcome; Test type: Other — A two-sided α-level of 0.05 will be used to determine the statistical significance; p = 0.1695, ANCOVA — Testing whether group means are different; A p-value < 0.05 indicates real discontinuation mean and sham discontinuation mean are different. Analyses adjusted for gender and baseline value; Difference in Group Means = -12.0, 95% CI 2-sided [-29.3 to 5.3] — Differences reported as the sham discontinuation mean minus the real discontinuation mean. These differences have been adjusted for gender and baseline total cholesterol value
Statistical Analysis 2: Comparison: Levothyroxine Group ("Sham Discontinuation") vs Placebo Group ("Real Discontinuation"); Analysis of 6-month LDL outcome; Test type: Other — A two-sided α-level of 0.05 will be used to determine the statistical significance; p = 0.3805, ANCOVA — Testing whether group means are different; [statistical method as in outcome 7, analysis 1]; Difference in Group Means = -6.8, 95% CI 2-sided [-22.2 to 8.6] — Differences reported as the sham discontinuation mean minus the real discontinuation mean. These differences have been adjusted for gender and baseline LDL values
Statistical Analysis 3: Comparison: Levothyroxine Group ("Sham Discontinuation") vs Placebo Group ("Real Discontinuation"); Analysis of 6-month HDL outcome; Test type: Other — A two-sided α-level of 0.05 will be used to determine the statistical significance; p = 0.5724, ANCOVA — Testing whether group means are different; [statistical method as in outcome 7, analysis 1]; Difference in Group Means = 1.7, 95% CI 2-sided [-4.44 to 7.9] — Differences reported as the sham discontinuation mean minus the real discontinuation mean. These differences have been adjusted for gender and baseline HDL values
Statistical Analysis 4: Comparison: Levothyroxine Group ("Sham Discontinuation") vs Placebo Group ("Real Discontinuation"); Analysis of 6-month triglyceride outcome; Test type: Other — A two-sided α-level of 0.05 will be used to determine the statistical significance; p = 0.3939, ANCOVA — Testing whether group means are different; [statistical method as in outcome 7, analysis 1]; Difference in Group Means = -17.8, 95% CI 2-sided [-59.4 to 23.9] — Differences reported as the sham discontinuation mean minus the real discontinuation mean. These differences have been adjusted for gender and baseline triglyceride values

ADVERSE EVENTS:
Time Frame: 6 months
Description: Of the 50 randomized participants, 24 were assigned to the LT4 group and 26 were assigned to the placebo group. There were 5 post-randomization exclusions, resulting in 21 participants in the LT4 group and 24 participants in the placebo group. One participant in the placebo group was discontinued (participant choice) prior to Week 6. This resulted in 21 participants in the LT4 group and 23 participants in the placebo group for the final analysis cohort.
Arm/Group | Levothyroxine Group ("Sham Discontinuation") | Placebo Group ("Real Discontinuation")
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/23
Serious Adverse Events (participants affected / at risk) | 3/21 | 1/23
Other Adverse Events (participants affected / at risk) | 9/21 | 15/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levothyroxine Group ("Sham Discontinuation") (N=21) | Placebo Group ("Real Discontinuation") (N=23)
Gangrene of toe (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
catheter ablation of arrhythmogenic focus (Cardiac disorders) | 1 (1) | 0 (0)
revision posterior decompression cervical cord and fusion (Surgical and medical procedures) | 1 (1) | 0 (0)
transurethral prostatectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
metastatic adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
fluoroscopy guided percutaneous insertion of drug eluting stent into coronary artery with contrast (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levothyroxine Group ("Sham Discontinuation") (N=21) | Placebo Group ("Real Discontinuation") (N=23)
fracture of rib (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Fractures
angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
cardiac pacemaker replaced (Cardiac disorders) | 0 (0) | 1 (1)
cellulitis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2)
cut of foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
cut of hand (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
dental restoration (Surgical and medical procedures) | 0 (0) | 1 (1)
dizziness (Nervous system disorders) | 0 (0) | 3 (3)
dry eye (Eye disorders) | 0 (0) | 1 (1)
fatigue (General disorders) | 0 (0) | 2 (3)
fluttering heart (Cardiac disorders) | 0 (0) | 1 (1)
fracture of phalanx of foot (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 0 (0) | 1 (2)
hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)
feels hot (Vascular disorders) | 0 (0) | 1 (1)
menopausal flushing (Vascular disorders) | 0 (0) | 1 (1)
hypertensive disorder (Vascular disorders) | 1 (1) | 0 (0)
bronchitis (Infections and infestations) | 1 (1) | 0 (0)
injection of knee (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
injury of lower leg (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
intravitreal injection of anti-vascular endothelial growth factor (Eye disorders) | 1 (1) | 0 (0)
kidney stone (Renal and urinary disorders) | 0 (0) | 1 (1)
labored breathing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
low blood pressure (Vascular disorders) | 1 (1) | 1 (1)
nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
carcinoma of prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
numbness of hand (Nervous system disorders) | 0 (0) | 1 (2)
open wound of buttock (Infections and infestations) | 0 (0) | 1 (1)
open wound of hip region (Infections and infestations) | 0 (0) | 1 (1)
injury of elbow (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
pain in coccyx (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
paresthesia of upper limb (Nervous system disorders) | 1 (1) | 0 (0)
removal of sebaceous cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
restenosis (Cardiac disorders) | 1 (1) | 0 (0)
scalp itchy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
shoulder pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
simple extraction of tooth (Surgical and medical procedures) | 1 (1) | 0 (0)
spasm (Nervous system disorders) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
lightheadedness (General disorders) | 0 (0) | 1 (1)
multiple joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
fall on ice (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
fractured dental restoration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
fixed prosthodontic procedure (Surgical and medical procedures) | 0 (0) | 1 (1)
polyp of sigmoid colon (Gastrointestinal disorders) | 1 (1) | 0 (0)
polyp of transverse colon (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-30): https://cdn.clinicaltrials.gov/large-docs/15/NCT04288115/Prot_SAP_001.pdf
  • Informed Consent Form (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT04288115/ICF_000.pdf